CLINICAL TRIAL: NCT01115985
Title: ASP1585 Pharmacokinetic Interaction Study - Pharmacokinetic Interaction With Atorvastatin -
Brief Title: A Study to Assess the Effect of ASP1585 on Pharmacokinetics of Atorvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1585-CL-0010
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Healthy; Pharmacokinetics of Atorvastatin
Keywords: ASP1585; Drug-drug interaction; Atorvastatin; Healthy volunteer
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single-add first group (Experimental): single administration first, then concomitant administration
  Interventions: Drug: ASP1585; Drug: atorvastatin
- combi-add first group (Experimental): concomitant administration first, then single administration
  Interventions: Drug: ASP1585; Drug: atorvastatin

INTERVENTIONS:
Drug: ASP1585 — oral
Drug: atorvastatin — oral
  Other Names: Lipitor

SUMMARY:
This study is to assess the effect of ASP1585 on pharmacokinetics of atorvastatin in 2x2 crossover method.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: =<50.0kg, <80.0kg
* Body mass index: =<17.6, <26.4
* Healthy as judged by investigator or caregiver from subjective and objective symptoms and physical examination data

Exclusion Criteria:

* Attending another clinical trial within 120 days before the study
* Blood donation within 90 days (400ml) or 30 days (200ml) before the study
* Receiving any drugs within 7 days before the study
* History of allergy to drugs
* Having GI disorders
* History or complication of liver diseases
* History or complication of heart disease
* History or complication of respiratory diseases
* History or complication of renal diseases
* History or complication of cerebrovascular diseases

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of atorvastatin | 48 hours after administration

SECONDARY OUTCOMES:
Safety assessed by AE, vital signs 12-lead ECG and lab tests | 7 days after administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Tokyo, Japan